CLINICAL TRIAL: NCT03802097
Title: Multicenter Randomized Controlled Trial About no Antimicrobial Prophylaxis for Patients Undergoing Totally Laparoscopic Distal Gastrectomy for Gastric Carcinoma (KSWEET-03)
Brief Title: Study About no Antimicrobial Prophylaxis in Totally Laparoscopic Distal Gastrectomy
Acronym: KSWEET-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean South West East Gastric Surgery Group (Other)
Responsible Party: Principal Investigator, Oh Jeong, MD, PhD, FACS, Korean South West East Gastric Surgery Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSWEET-03
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer; Complication of Surgical Procedure
Keywords: Gastric cancer; Laparoscopic gastrectomy; Prophylactic antibiotics; Infectious complications
MeSH Terms: conditions — Stomach Neoplasms | interventions — Adenosine Monophosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (treatment group) (Experimental): No use of antimicrobial prophylaxis
  Interventions: Procedure: No use of antimicrobial prophylaxis
- B group (control group) (Experimental): Use of antimicrobial prophylaxis
  Interventions: Procedure: Use of antimicrobial prophylaxis

INTERVENTIONS:
Procedure: No use of antimicrobial prophylaxis — Do not use of prophylactic antimicrobial for the patients with undergoing totally laparoscopic distal gastrectomy with D1 or D1+ lymphadenectomy for the gastric cancer
  Other Names: No AMP
  Arms: A group (treatment group)
Procedure: Use of antimicrobial prophylaxis — Use of prophylactic antimicrobial for the patients with undergoing totally laparoscopic distal gastrectomy with D1 or D1+ lymphadenectomy for the gastric cancer
  Other Names: AMP
  Arms: B group (control group)

SUMMARY:
Laparoscopic gastrectomy has fewer infectious complications compared to open surgery. Recently, the incidence of postoperative infectious complications was greatly reduced due to the development of surgical techniques and improvement of prevention and control of surgical infection. Previous multicenter, phase II study (KSWEET-01) revealed that the incidence of infectious complications of laparoscopic gastrectomy without prophylactic antibiotics was not significantly higher than previously reported data.

Therefore, this study aim to prove the safety of totally laparoscopic distal gastrectomy without prophylactic antibiotics, specially reference to the postoperative infectious complications.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the non-inferiority of incidence of infectious complications in the experimental group that did not use prophylactic antibiotics compared to the control group using prophylactic antibiotics.

The primary endpoint is the incidence of surgical site infections within 30 days after surgery and the difference limit of the non-inferiority of the experimental group is assumed to be - 0.05 (5%). Assuming that the incidence of postoperative infectious complications in the control group is 5% and the incidence of infectious complications in the experimental group is assumed to be about 8%. It is assumed that the significant level is 5% and the power is at least 80%.

According to the above method, a total of 260 patients (130 patients in each group) are needed when 117 patients are needed in each group and about 10% of drop rates and protocol violence are considered.

ELIGIBILITY:
Inclusion Criteria:

* A patient undergoing totally laparoscopic distal gastrectomy for the gastric cancer located in the low or middle part of the stomach
* A patient who underwent limited lymphadenectomy (D1 or D1+) with clinical T1-2N0M0 stage based on 8th edition of the International Union Against Cancer (UICC) tumor node metastasis (TNM) classification
* From 18 to 75 years old
* Eastern Cooperative Oncology Group (ECOG) status 0-1
* American Society of Anesthesiologists (ASA) score I-II
* A patient with appropriate bone marrow function, renal function, lung function, and liver function
* Before the surgery, decide to participate in this study and agree with the written informed consent

Exclusion Criteria:

* A patient who underwent previous abdominal surgery
* Combined other abdominal organ cancer
* A patient who received chemotherapy and radiotherapy within the last 6 months
* Combined organ resection other than cholecystectomy
* A patient undergoing emergency surgery due to perforation or bleeding
* A patient who have received antibiotic treatment for other infectious diseases within one month of operation
* Severely malnourished patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infections within 30 days | within 30 days after operation
  The diagnosis of infectious complications is made according to the Centers for Disease Control and Prevention (CDC) surgical site infection diagnosis criteria according to physical or radiological findings.

SECONDARY OUTCOMES:
Length of hospital stay | up to 6 months
  From date of operation until the date of hospital discharge
Incidence of remote non-surgical site infections | within 30 days after operation
  Any postoperative infectious complications other than surgical site infections

CONTACTS AND LOCATIONS:
Overall Officials: Oh Jeong, M.D.,Ph.D., Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jellanamdo, South Korea

IPD SHARING:
Plan to Share IPD: No